CLINICAL TRIAL: NCT06097000
Title: A Study of the Safety and Efficacy of Intelligent Powered Exoskeletons in Postoperative Spinal Rehabilitation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: BEIJING DNSYS INNOVATION Co. Ltd (Unknown); Beijing Haidian Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XW-NS-IPEPSR
Record Dates: First submitted 2023-09-27; First posted 2023-10-24 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Exoskeleton Device
Keywords: Hip Exoskeleton Device; Spinal Cord Injuries; Rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Powered Exoskeleton Group (Experimental): Rehabilitation exercises with powered exoskeletons
  Interventions: Device: powered exoskeletons
- Traditional Group (No Intervention): Rehabilitation exercises without the use of powered exoskeletons

INTERVENTIONS:
Device: powered exoskeletons — Whether to use powered exoskeletons for exercise rehabilitation
  Arms: Powered Exoskeleton Group

SUMMARY:
Systematic and professional rehabilitation training is generally effective for patients with lower limb dyskinesia, but most of them lose the chance of recovery due to failure to receive systematic rehabilitation treatment. Our team has developed an intelligent power armor for patients with lower limb motor dysfunction, which can assist patients to complete high-quality rehabilitation training. In order to evaluate the safety and efficacy of the Smart Power Armor for post-surgical spine patients, and to provide data support for a confirmatory clinical study, we designed a single-center, prospective, randomized controlled study to compare the level of recovery of lower limb motor function in patients with different rehabilitation strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old;
* Spinal surgery within 1 year due to degeneration, tumor, trauma or other reasons, postoperative motor disorders of both lower limbs, such as muscle weakness (3-5 level reduction), increased muscle tone, gait incoordination caused by deep sensory loss, etc.;
* The patient does not have a plan to rehabilitate in a specialized rehabilitation hospital, and plans to rehabilitate at home;

Exclusion Criteria:

* Short expected survival from malignant diseases;
* Muscle strength is less than grade 3, and the muscles of both lower limbs are severely atrophied;
* Suffering from other neurological diseases;
* Planned to undergo other surgeries within 3 months;
* Unable to cooperate with the transmission power external armor or cooperate with the rehabilitation training due to the physical condition;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test | 3 months
  meter; distance participants walked as fast as possible in a flat corridor in six minutes

SECONDARY OUTCOMES:
Average rate of change in muscle strength | 3 months
  (change in muscle strength level* number of persons)/total number of persons enrolled in the group
10 meter autonomous walking test | 3 months
  meter; participants walk ten meters at a self-selected speed
10 meter fast walking test | 3 months
  meter; participants walk ten meters at fastest speed
rate of change in hip joint mobility | 3 months
  (hip joint mobility with assistance - hip joint mobility without assistance)/hip joint mobility without assistance; use joint mobility scales to measure hip joint mobility
stride length | 3 months
  centimeter; left and right legs are measured separately
rate of change in heart rate | 3 months
  (post-training heart rate - resting heart rate)/resting heart rate
rate of change in arterial partial pressure of oxygen | 3 months
  (post-training arterial partial pressure of oxygen - arterial partial pressure of oxygen at rest)/arterial partial pressure of oxygen at rest
adverse event incidence rate | 12 months
  Number of cases of adverse events/number of enrollees
serious adverse event incidence rate | 12 months
  Number of cases of serious adverse events/number of enrollees
Thigh Swing Speed | 3 months
  degrees/second; left and right legs are measured separately
Thigh Lifting Moment | 3 months
  Newton*Meter; left and right legs are measured separately
Thigh Swing Angle | 3 months
  degree; left and right legs are measured separately

CONTACTS AND LOCATIONS:
Locations (1):
- Intelligent Powered Exoskeleton, Beijing, Beijing Municipality, China